CLINICAL TRIAL: NCT05101668
Title: A Prospective, Multi-center, Single-arm Objective Performance Criteria Trial to Evaluate the Safety and Efficacy of Intracranial Thrombus Aspiration Catheter in Treatment of Acute Large-vessel Occlusive Stroke
Brief Title: Safety and Efficacy of Intracranial Thrombus Aspiration Catheter in the Treatment of Acute Large-vessel Occlusive Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: According to the Medical Device Classification Catalogue issued by the NMPA in 2022, the registration path of intracranial aspiration catheter is clinical evaluation, and clinical trials are not required.
Sponsor: Sinomed Neurovita Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SINOMED ADPAT
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Aspiration; Acute Ischemic Stroke; Large-vessel Occlusion
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, single-arm objective performance criteria
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intracranial Thrombosis Aspiration Catheter (Experimental): Intracranial Thrombosis Aspiration Catheter, product of Sinomed Neurovita Technology Inc.
  Interventions: Device: Intracranial Thrombosis Aspiration Catheter

INTERVENTIONS:
Device: Intracranial Thrombosis Aspiration Catheter — Direct Aspiration

SUMMARY:
A prospective, multicenter, single-arm objective performance criteria trial to investigate the safety and efficacy of SINOMED ADPAT for Recanalization Therapy in acute large-vessel occlusive stroke.

DETAILED DESCRIPTION:
This study plans to recruit 164 patients with acute intracranial large-vessel occlusion within 24 hours time window. The Primary endpoint is the instant recanalization rate of target vessel after operation. Secondary efficacy endpoints will include: 1) immediate recanalization rate of the first pass of aspiration; 2) the recanalization time of the target vessel blood flow; 3) the improvement of the postoperative NIHSS score; 4) the ratio of good neurological function (mRS 0-2 points) at 90 days; 5) the success rate of device; 6) the success rate of operation; 7) The proportion of rescue therapy. Safety endpoints will include: 1) the incidence of symptomatic intracranial hemorrhage within 24 hours after operation; 2) all-cause death and stroke-related mortality at 90 days; 3) stroke recurrence rate within 90 days after operation; 4) surgery-related complications; 5) adverse events; 6) serious adverse events; 7) Device defection rate

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years and ≤ 85 years;
2. Acute ischemic stroke, patients with anterior / posterior circulation vessel occlusion (intracranial segment of internal carotid artery or M1 or M2 segment of middle cerebral artery) confirmed by digital subtraction angiography (DSA);
3. Premorbid modified Rankin Scale(mRS)<2 and Pre-operation NIHSS score ≥6;
4. The patients should receive endovascular treatment within 24 hours:

   1. If the treatment could happen within 6 hours, the patient should have an CT or MR
   2. If the treatment could happen 6-24 hours, the patient should have an CT or magnetic resonance (MR), have an ASPECTS ≥ 6 points. If immediate CT perfusion imaging or MR perfusion imaging is feasible, CT perfusion (CTP) or magnetic resonance perfusion (MRP) should be performed at the same time to assist in the evaluation of the infarct core.
5. Written informed consent obtained from patient or patient's legally authorized representative.

Exclusion Criteria:

1. Large (more than one-third of the MCA) regions of clear hypodensity on the baseline neuroimaging or significant mass effect with midline shift;
2. Any type of intracranial hemorrhage or subarachnoid hemorrhage (only microbleeds are allowed, or judge from surgeon's clinical experience) by neuroimaging;
3. Proven Simultaneous acute occlusion of both carotid artery systems, and Proven tandem lesion of simultaneous occlusion of intracranial and extracranial vessels by neuroimaging;
4. Occlusion of the common carotid artery,and known or suspected chronic occlusion of target vessel;
5. Patients with consciousness disorder with posterior circulation vascular occlusion, NIHSS score is 3 points (1a=3);
6. Proven intracranial artery occlusion due to arterial dissection or arteritis by neuroimaging;
7. Arterial tortuosity and other problems that would prevent the device from reaching the target vessel;
8. Known to have one or more of the following allergies/resistances or contraindications: antiplatelet drugs/anticoagulant drugs/contrast agents and/or anesthetics;
9. Known allergies to medical devices and related products (allergy to materials such as nickel-titanium metal or its alloys);
10. Active bleeding or known bleeding tendency (such as: anticoagulant therapy or coagulation dysfunction before surgery, international normalized ratio (INR)>3.0);
11. Baseline platelet counts<40×10^9/L;
12. Severe heart, liver or kidney failure and other serious or terminal illness;
13. Accompanied by ST-segment elevation myocardial infarction or severe infection (endocarditis or sepsis);
14. Hypertension that cannot be controlled after treatment (Baseline blood pressure>185/110 mmHg);
15. Baseline blood glucose < 2.7 or > 22.2 mmol/L. after treatment;
16. Life expectancy less than 3 months;
17. Women who are pregnant or planning to pregnancy during half a year by taking medical history);
18. Dementia or psychiatric disease that would confound the neurological or functional evaluations;
19. Current participation in another drug or device research;
20. Other special situations which the researchers believe to be not suitable for enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Instant recanalization rate of target vessel after operation | Last aspiration
  Instant recanalization rate (mTICI 2b-3) of target vessel after operation

SECONDARY OUTCOMES:
Instant recanalization rate of target vessel after the first aspiration | First aspiration
  Instant recanalization rate (mTICI 2b-3) of target vessel after the first aspiration
The recanalization time of the target vessel blood flow | Procedure time (femoral artery puncture to recanalization)
  The recanalization (mTICI 2b-3) time of the target vessel blood flow
The improvement of the postoperative NIHSS score the improvement of the postoperative NIHSS score | Change in NIHSS score at preoperative、24(-6/+24) hours、7±2 days or discharge
  NIH Stroke Scale/Score (NIHSS)：Calculates the NIH Stroke Scale for quantifying stroke severity.
Proportion of good neurological function (mRS 0-2) | 90 days
  The modified Rankin Scale/Score (mRS) : scores of 0 to 2 were defined as good neurological function (treatment success)
The success rate of device | Intraoperative
  The intracranial thrombus aspiration catheter was successfully delivered to the occluded segment of the blood vessel and then successfully released, and suction was performed, and the delivery system was successfully withdrawn.
The success rate of operation | End of Procedure
  The success of recanalization after the final treatment (mTICI 2b-3, allowing the use of rescue therapy)
The incidence of symptomatic intracranial hemorrhage | 24(-6/+24) hours
  Through Heidelberg Bleeding Classification to evaluate the intracranial hemorrhage (National Institutes of Health Stroke Scale (NIHSS) score of ≥4 points)
All-cause death and stroke-related mortality | 90 days
  All-cause death and stroke-related mortality
The rate of Stroke recurrence | 90 days
  The existence of clear imaging evidence to confirm that the target vessel is occluded again, which leads to an ischemic stroke event.
Procedure-related complications | Intraoperative
  Procedure-related complications: including arterial rupture, arterial dissection, distal thromboembolism, vascular puncture site complications, etc
Adverse events and serious adverse events | During the clinical trials
  Any adverse events and serious adverse events are associated with clinical trials in human
The rate of device defection | Intraoperative
  Device defection

CONTACTS AND LOCATIONS:
Overall Officials: Qingwu Yang, M.D/Ph.D, Principal Investigator — The Second Affiliated Hospital of Army Medical University; Yimin Liu, M.D/Ph.D, Principal Investigator — Wuhan University
Locations (6):
- China (6):
  - Qingwu Yang, Chongqing
  - LIUZHOU People's Hospital, Liuchow
  - Jinzhao Liu, Pujiang
  - Zhongnan Hospital of Wuhan University, Wuhan
  - Xiangtan Central Hospital, Xiangtan
  - Xiang Yang No.1 Peoples Hospital, Xiangyang